CLINICAL TRIAL: NCT00626899
Title: Comparison of the Performance of a New Pulse-contour Analysis Cardiac Output Measurement (Vigileo) With the Traditional Method in Patients With Induced Therapeutic Hypothermia After Cardiac Arrest
Brief Title: Comparison Performance Vigileo vs. Continuous CCO (Vigilance) in Patients With Induced Therapeutic Hypothermia
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Matthias Haenggi, Department of Intensive Care Medicine, University Hospital Bern - Inselspital
Other Study IDs: KIM-Vig/Vig
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Cardiac Arrest; Hypothermia, Induced
Keywords: Validation of Cardiac Output measurement in hypothermic patients
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients resuscitated from a cardiac arrest undergo therapeutic hypothermia as a treatment option. Measuring the cardiac output in these patients is sometimes important, but difficult, as these patients require an invasive device for measurement. Recently, a non-invasive device based on pulse-contour analysis of the arterial pulse was developed (the Vigileo). Hypothermia changes the pulse contour, so the performance of the Vigileo in patients with induced therapeutic hypothermia is not known. Therefore we conduct this observational study in which the cardiac output of the patients is measured with the traditional method and the Vigileo simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* patients who survived a cardiac arrest and are treated with therapeutic hypothermia
* pulmonary arterial catheter placed by treating physician

Exclusion Criteria:

* arterial catheter placement is contraindicated
* Aortic valve insufficiency (moderate to severe)
* placement of intra-aortic balloon pump (IABP) or a LVAD (left ventricular assist device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac arrest who are treated with therapeutic hypothermia and require a PAC for hemodynamic monitoring
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Haenggi, MD, Principal Investigator — Departement of Intensive Care Medicine, University Hospital Bern, Inselspital, Bern, Switzerland
Locations (1):
- Departement of Intensive Care Medicine - University Hospital Bern - Inselspital, Bern, Switzerland